CLINICAL TRIAL: NCT04089657
Title: Apatinib Plus Sintilimab in Patients With Advanced Gastric Cancer
Brief Title: Apatinib Plus Sintilimab in Advanced Gastric Cancer Refractory to at Least Two Previous Chemotherapy Regimens
Acronym: ASGARD
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fujian Cancer Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: APAICI
Record Dates: First submitted 2019-09-10; First posted 2019-09-13 (Actual); Last update posted 2019-09-13 (Actual); Status verified 2019-09

CONDITIONS: Advanced Metastatic Gastric Cancer
MeSH Terms: interventions — apatinib; sintilimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Apatinib+Sintilimab (Experimental): Apatinib 500mg qd p.o and Sintilimab 200mg intravenously on day 1 every 3 weeks until disease progression or intolerable toxicity or patients withdrawal of consent
  Interventions: Drug: Apatinib Mesylate; Drug: Sintilimab

INTERVENTIONS:
Drug: Apatinib Mesylate — Apatinib 500mg qd, oral, taken half an hour after a meal
  Other Names: Apatinib
Drug: Sintilimab — Sintilimab 200mg intravenously on day 1
  Other Names: IBI308

SUMMARY:
The purpose of this study is to assess the efficacy and safety of Apatinib combined with PD-1 antibody Sintilimab for for Chemotherapy-Refractory Advanced Metastatic Gastric Cancer

DETAILED DESCRIPTION:
Patients with advanced gastric cancer (AGC) can be treated with multiple lines of chemotherapy. After second-line treatment some patients may receive third- and subsequent lines of chemotherapy if their performance status is well-preserved and they are willing to receive subsequent active treatments. Apatinib is a small-molecule VEGFR-2 tyrosine kinase inhibitor approved by the CFDA for the treatment of advanced gastric cancer. In a phase III trial, apatinib significantly improved PFS and OS compared with placebo, but the clinical benefit was modest. As a result of toxicity, 850 mg/day Apatinib may cause dose reduction and delay in some patients ,which also caused some doubts. Therefore, it is a reasonable treatment strategy by reducing the dose and combining it with another low-toxic drug to achieve similar or better effects. Some studies have shown that the combination of targeted therapy and immunotherapy may be effective in solid tumor. Sintilimab (IBI308) is a monoclonal antibody targeting programmed death-1 (PD-1). So, the investigators designed an open-label, single-arm, phase II clinical study to evaluate the efficacy and safety of apatinib combined with Sintilimab in Chemotherapy-Refractory Advanced Metastatic Gastric Cancer.

ELIGIBILITY:
Inclusion Criteria:

* Age between 20-75 years old
* Has histologically confirmed diagnosis of unresectable locally advanced,recurrent or metastatic gastric or GEJ adenocarcinoma
* Life expectancy of more than 3 months
* Eastern Cooperative Oncology Group (ECOG) performance status was 0 - 1
* Have failed for at least 2 lines of chemotherapy
* At least 3 weeks from previous chemotherapy at first dose of trial drug
* Resolution of all acute toxic side effects of prior therapy or surgical procedures to grade ≤ 1 National Cancer Institute-Common Toxicity Criteria (NCI-CTC) (except for the laboratory values)
* Failure of prior palliative chemotherapy/chemotherapies (at least one irinotecan- or cisplatin-based). Failure is defined either by progression of disease or by significant toxicity that precludes further treatment.
* At least one measurable lesion defined by RECIST 1.1 as determined by investigator assessment.
* Has adequate organ function
* At least 4 weeks from any major surgery (at first dose of trial drug)
* Patients must be able to swallow apatinib

Exclusion Criteria:

* In the past, participants have received anti PD-1, anti PD-L1 or anti PD-L2 drugs or drugs targeting another stimulation or synergistic inhibition of T cell receptors (such as Cytotoxic T-Lymphocyte Antigen 4 [CTLA-4] and CD137)
* Other co-existing malignancies or malignancies diagnosed within the last 5 years(except cured cutaneum carcinoma or carcinoma in situs of cervix)
* Less than 4 weeks from the last clinical trial
* Active and uncontrollable bleeding from gastrointestinal tract
* Known history of QT interval prolongation, ongoing QT prolongation (> 450 msec for males or > 470 msec for females), any cardiac ventricular dysrhythmias, atrial fibrillation of any grade
* Hypertension that cannot be controlled by medications (> 140/90 mmHg despite optimal medical therapy)
* Abnormal Coagulation (INR>1.5、APTT>1.5 UNL), with tendency of bleed;
* Factors that could have an effect on oral medication (such as inability to swallow, chronic diarrhea and intestinal obstruction);
* Active uncontrolled infection
* Known human immunodeficiency virus (HIV) infection
* Symptomatic central nervous metastasis and/or cancerous meningitis
* Known allergic/hypersensitivity reaction to any of the components of the treatment; or known drug abuse/alcohol abuse
* Pregnant or lactating women

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-12-01 (Estimated); Primary Completion 2020-12-01 (Estimated); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
Disease control rate(DCR) | 12 months
  The percentage of patients who have achieved complete response, partial response and stable disease,evaluated by RECIST, confirmed at least 4 weeks following the date of the initial response.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | 12 months
  The percentage of patients who achieve complete response or partial response,evaluated by RECIST, confirmed at least 4 weeks following the date of the initial response.
Overall survival (OS) | up to 12 months
  Overall survival (OS) was calculated from the date of initial treatment with apatinib to the date of death due to any cause.
Duration of Response (DOR) | up to 12 months
  Time from date of first RECIST response to progressive disease [PD] or death
Progression Free Survival (PFS) | up to 12 months
  PFS was calculated from the day of randomization to the date of first documented progression, or death from any cause.
Adverse events（AE） | up to 12 months
  Adverse events assessed using the NCI common toxicity criteria, version 4.01

CONTACTS AND LOCATIONS:
Overall Officials: Nanfeng Fan, MD, Study Chair — Fujian Cancer Hospital

IPD SHARING:
Plan to Share IPD: No